CLINICAL TRIAL: NCT07369830
Title: The Impact of Probiotic Intervention on the Gut Microbiota and Bowel Function of Patients With Prophylactic Ileostomy for Ultra Low Rectal Cancer -a Multicenter Randomized Controlled Trial
Brief Title: The Impact of Probiotic Intervention on the Gut Microbiota and Bowel Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: Characteristic Medical Center of Rocket Army (Unknown); Zhongnan Hospital (Other); The First Affiliated Hospital of Nankai University (Unknown); First Affiliated Hospital of Fujian Medical University (Other); Ruijin Hospital (Other); Nanfang Hospital, Southern Medical Universit (Unknown)
Responsible Party: Principal Investigator, Jianbin Xiang, Principal Investigator, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-1273
Record Dates: First submitted 2025-12-23; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; intersphincteric resection; prophylactic ileostomy; probiotic intervention; bowel function
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The low dose group received interventions (4 Meiya pills, administered into the dysfunctional intestine once a week) starting 1 week after the ileostomy the high dose group received interventions (4 Meiya pills, administered into the dysfunctional intestine twice a week) starting 1 week after the ileostomy the control group received routine postoperative follow-up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high dose group (Experimental): the high dose group received interventions (4 Clostridium butyricum (live) Tablets(Meiya), administered into the dysfunctional intestine twice a week) starting 1 week after the ileostomy
  Interventions: Biological: Clostridium butyricum (live) Tablets(Meiya)
- low dose group (Experimental): the low dose group received interventions (4 Clostridium butyricum (live) Tablets(Meiya), administered into the dysfunctional intestine once a week) starting 1 week after the ileostomy
  Interventions: Biological: Clostridium butyricum (live) Tablets(Meiya)
- control group (No Intervention): the control group received routine postoperative follow-up

INTERVENTIONS:
Biological: Clostridium butyricum (live) Tablets(Meiya) — Clostridium butyricum (live) Tablet administered into the dysfunctional intestine for low dose and high dose group, while control group has no intervention
  Arms: high dose group; low dose group

SUMMARY:
This study aims to propose a novel, easy-to-operate intervention strategy that effectively improves defecation function after stoma reversal and to assess its impact on the gut microbiota.The efficacy and safety of antegrade placement of probiotics into the distal deserted intestine during prophylactic stoma to improve bowel function after stoma reversal were evaluated through randomized controlled clinical trials.Observing the changes in gut microbiota during the prophylactic stoma period, the impact of probiotics on the structure of gut microbiota, and exploring the correlation between gut genera and bowel function after stoma reversal.

DETAILED DESCRIPTION:
This study includes patients with ultra low rectal cancer who underwent ISR（Intersphincteric Resection） and prophylactic ileostomy. Patients are randomly assigned to the low dose group,high dose group and the control group in a 1:1:1 ratio. The low dose group received interventions (4 Meiya pills, administered into the dysfunctional intestine once a week) starting 1 week after the ileostomy, the high dose group received interventions (4 Meiya pills, administered into the dysfunctional intestine twice a week) starting 1 week after the ileostomy, while the control group received routine postoperative follow-up. Evaluation indicators included bowel function and quality of life before the prophylactic ileostomy and 1 week, 2 weeks, 1 month, 3 months, and 6 months and so on until two years after the stoma reversal.

Fecal samples are collected prior to prophylactic ileostomy. Post-stoma reversal surgery, fecal samples are obtained from patients at their first defecation . All fecal samples underwent 16s rRNA gene sequencing and bioinformatic analysis to compare the microbial composition differences among three groups. Key genera associated with bowel function were identified through correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years
2. Ultra low rectal cancer meeting the indication for Intersphincteric Resection (ISR) surgery
3. Underwent a prophylactic ileostomy
4. Scheduled for stoma reversal surgery within 6 months after the ISR procedure
5. Digestive tract reconstruction achieved via either hand-sewn or stapled coloanal anastomosis
6. Patient has a strong preference for undergoing sphincter-preserving surgery
7. Capable of understanding and willing to provide signed informed consent

Exclusion Criteria:

1. Does not meet the surgical indications for Intersphincteric Resection (ISR)
2. Presence of multiple primary colorectal malignancies
3. Patients who have received neoadjuvant radiotherapy
4. Patients who experience disease progression or death in the postoperative period
5. Patients who develop severe anastomotic complications postoperatively, such as anastomotic leakage or stenosis
6. Patients whose actual stoma reversal surgery occurs more than 6 months after the ISR procedure
7. Patients who require long-term(more than 3 months) use of antibiotics
8. History of allergy to Clostridium butyricum (live) Tablets (MIYA) or any of its components
9. Concurrent use of other probiotic during the study period
10. Coexisting inflammatory bowel disease
11. History of neurological or psychiatric disorders, including but not limited to Parkinson's disease, Alzheimer's disease, organic brain diseases, stroke, epilepsy, or major psychiatric disorders (e.g., major depressive disorder)
12. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Low Anterior Resection Syndrome Score（LARS Score） | One month after stoma reversal
  Comparison of LARS scores among the three groups at one month postoperatively. Low Anterior Resection Syndrome (LARS) is characterized by major symptoms including difficulty defecating, urgency, incontinence of liquid stool, incontinence of flatus, and increased frequency of bowel movements. Based on severity, LARS can be classified as none (0-20 points), minor (21-29 points), or major (30-42 points) using LARS score. And higher scores mean a worse outcome.
microbial diversity | The first stool sample will be collected within one week before ISR surgery, and the second stool sample will be collected within three to five days after stoma reversal, upon the first bowel movement.
  Fecal samples from study participants with ISR preoperatively and postoperatively will be collected to analyze the alpha and beta diversity of gut microbiota among the three groups

SECONDARY OUTCOMES:
Wexner Incontinence Score | one month after ISR
  The Wexner Incontinence Score (WIS) assesses the severity of incontinence from five aspects: solid stool incontinence, liquid stool incontinence, flatus incontinence, pad usage, and lifestyle alterations. The score ranges from 0 to 20, where 0 represents normal and 20 represents complete incontinence.
Kirwan Incontinence Score | one month after ISR
  This grading system classifies anal incontinence into five grades (I-V) based on symptom severity: Grade I: No incontinence; Grade II: Incontinence to flatus or liquid stool; Grade III: Occasional solid stool incontinence; Grade IV: Frequent solid stool incontinence; Grade V: Requires a stoma (fecal diversion). Among these, Grades I-II indicate good continence function, while Grades III-IV indicate poor continence function.
Exploratory LARS Scoring Instrument | one month after ISR
  An exploratory scoring instrument was used to determine the severity of 16 specific variables that were identified by the Delphi consensus for defining LARS. In accordance with the response range defined by the WIS, there were 5 frequency options ranging from never (meaning no episodes; score 0) to always (meaning 1 or more episodes/day; score 4) for each item. Given that social and psychological features (marital separation, divorce, widowed seniors, etc) may have an influence on "relationships and intimacy," its response category for "never" was replaced with dichotomous options of "none" and "N/A." The summary score, also called the Delphi consensus severity score, was used as an index for patient-reported severity of LARS, ranging from 0 (best) to 64 (worst).
Fecal Incontinence Quality of Life (FIQL) Scale | one month after ISR
  The Fecal Incontinence Quality-of-Life (FIQL) Scale was used to analyze CSQoL. The FIQL entails 29 items that cover 4 domains: lifestyle (10 items), coping/behavior (9 items), depression/self-perception (7 items), and embarrassment (3 items).19 Each item has a range of 1 to 4 (except 2 items in depression/self-perception with ranges of 1-5 and 1-6). The score for each domain is the average of all items within its domain, and the global score is the mean of all domains. Higher scores indicate better CSQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Jianbin, Doctor, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this article (text, tables, figures, and appendices) will be shared. The study protocol, statistical analysis plan, and informed consent form will also be available. Data will be available beginning 9 months and ending 36 months after article publication. Proposals for data access should be directed to the corresponding author. To gain access, data requestors will need to sign a data access agreement. Data will be provided via a secure online platform.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 9 months and ending 36 months after article publication.
Access Criteria: De-identified individual participant data will be available to qualified researchers whose proposals have been approved by an independent data access committee. Requestors must submit a scientifically sound research proposal and sign a data use agreement.